CLINICAL TRIAL: NCT07245329
Title: Effect of Full-House Endoscopic Sinus Surgery With Versus Without Nasopharyngeal Lymphoid Ablation on Local Mucosal Inflammation in Chronic Rhinosinusitis With Nasal Polyps
Brief Title: Effect of Full-House ESS With Nasopharyngeal Lymphoid Tissue Ablation on Nasal Polyps
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Yin Yao, Professor of Otolaryngology-Head & Neck Surgery; Deputy Dean of Institute of Allergy and Clinical Immunology, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ-IRB202506055
Record Dates: First submitted 2025-09-21; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Nasal Polyps
Keywords: Full-House Endoscopic Sinus Surgery; Nasopharyngeal Lymphoid Tissue Ablation
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full-House Endoscopic Sinus Surgery Combined with Nasopharyngeal Lymphoid Tissue Ablation (Experimental)
  Interventions: Procedure: Nasopharyngeal Lymphoid Tissue Ablation; Procedure: Full-House Endoscopic Sinus Surgery
- Full-House Endoscopic Sinus Surgery (Active Comparator)
  Interventions: Procedure: Full-House Endoscopic Sinus Surgery

INTERVENTIONS:
Procedure: Nasopharyngeal Lymphoid Tissue Ablation — The nasal mucosa is initially decongested using a topical vasoconstrictor. A small-caliber urethral catheter is then introduced through each nasal cavity to elevate the soft palate. A 45° rigid nasoendoscope is inserted transorally to visualize the nasopharynx. Under endoscopic guidance, the nasopharyngeal lymphoid tissue is identified on the nasopharyngeal roof. Following aspiration of any secretions, the tissue is completely resected with a plasma scalpel.
  Arms: Full-House Endoscopic Sinus Surgery Combined with Nasopharyngeal Lymphoid Tissue Ablation
Procedure: Full-House Endoscopic Sinus Surgery — After complete removal of the nasal polyps, a full ethmoidectomy is performed, removing all bony septa within the sinuses. Conventional sphenoidotomy and frontal sinusotomy are carried out, with or without preservation of the middle turbinate. Only irreversibly polypoid mucosa is resected, while normal mucosa is preserved.

SUMMARY:
This study is designed to evaluate whether the addition of nasopharyngeal lymphoid tissue ablation to full-house endoscopic sinus surgery (ESS) provides superior control of nasal mucosa inflammation compared to full-house ESS alone in patients with nasal polyps. Thirty-two adult participants will be randomly assigned to undergo either full-house ESS only or full-house ESS combined with nasopharyngeal lymphoid tissue ablation. The primary outcome will be assessed through changes in inflammatory cell profiles at 1, 3, and 6 months postoperatively. Secondary outcomes include inflammatory cytokine levels, symptom scores, endoscopic findings, polyp recurrence rates, and safety measures.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Diagnosed with CRSwNP according to EPOS criteria
* Blood eosinophil count > 0.3 × 10⁹/L

Exclusion Criteria:

* Pregnant or lactating women.
* Cystic fibrosis
* primary ciliary dyskinesia
* fungal ball rhinosinusitis
* systemic vasculitis or granulomatous disease
* malignancy
* immunodeficiency.
* Subjects with an upper-respiratory-tract infection within the past 4 weeks.
* Clinically significant metabolic, cardiovascular, immune, neurologic, hematologic, gastrointestinal, cerebrovascular, or respiratory disorders, or any condition that, in the investigator's opinion, could interfere with outcome assessment or compromise patient safety.
* Currently participating in another clinical trial or having participated in one within 30 days, or staff directly involved in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Numbers and Proportions of Nasal Mucosa inflammatory cells in Patients With Nasal Polyps at Baseline and 1, 3, and 6 Months After Surgery | At baseline (before surgery) and 1 month, 3 months, and 6 months after surgery.
  Sampling of the ethmoid sinus mucosa from patients after surgery is performed under nasal endoscopic guidance; nasopharyngeal swabs are used to collect samples from the nasopharynx. The method for nasopharyngeal sampling is as follows: The subject sits in a seated position, blows their nose, and closes their eyes before swab sample collection to facilitate relaxation and ease of sampling. A professional doctor gently inserts the nasal swab into one nostril along the bottom of the nasal cavity (parallel to the hard palate) until it reaches the nasopharynx, then rotates the swab approximately five times in the nasopharynx. The swab is placed into a collection tube containing 2 mL of RPMI medium. One nasopharyngeal swab is collected per donor each time. After processing, flow cytometry is used for analysing the numbers and proportions of inflammatory cells (including T cells, B cells, Plasma cells, Eosinophils, and Neutrophils).

SECONDARY OUTCOMES:
Inflammatory Cytokine Levels in Nasal Secretions Post - surgery | At baseline (before surgery) and 1 month, 3 months, and 6 months after surgery.
  Detection of inflammatory cytokine levels (e.g., IL - 5, IL - 13) in nasal secretions. Samples are collected via nasal swab, then processed and analyzed using immunoassay techniques (e.g., ELISA).
Total VAS Score and Symptom - specific VAS Scores Post - surgery | At baseline (before surgery) and 1 month, 3 months, and 6 months after surgery.
  Evaluate total VAS score and individual symptoms (nasal obstruction, mucopurulent discharge, postnasal drip, headache/dizziness, facial fullness, hyposmia/anosmia, sneezing, sleep disturbance, fatigue, general discomfort). Scores are self - reported by patients using a 0 - 10 scale.
Nasal Endoscopy Scores | At baseline (before surgery) and 1 month, 3 months, and 6 months after surgery.
  Assess nasal endoscopy scores. The scoring includes signs such as nasal polyps, mucosal edema, secretions, crusting, and scarring. Trained clinicians perform nasal endoscopy at each time point following a standardized protocol and record scores based on the presence and severity of these signs.
SNOT - 22 Score Changes Post - surgery | At baseline (before surgery) and 1 month, 3 months, and 6 months after surgery.
  Assess quality - of - life symptoms (nasal discharge, sneezing, rhinorrhea, cough, postnasal drip, purulent discharge, smell/taste disturbance, nasal obstruction/congestion, ear fullness, dizziness, ear pain, facial pain/pressure, difficulty falling asleep, nighttime awakenings, poor sleep quality, morning fatigue, daytime fatigue, decreased work efficiency, difficulty concentrating, depression/irritability, anxiety, restlessness) via the SNOT - 22 questionnaire.
Polyp Recurrence Post-surgery | Focus on the first 6 months post-surgery, with extended monitoring continuing up to 24 months.
  Polyp recurrence assessed by nasal endoscopy.
Rate of Reoperation | Focused on 6 months post-surgery; continued monitoring to 24 months post-surgery.
  Assess the proportion of patients undergoing reoperation within 6 months after surgery. Reoperation is indicated if:
  * Oral methylprednisolone (>2 courses: 3 - week tapering, initial dose 30 mg) fails to control mucosal edema/inflammation (polyp score ≥2) and severe nasal symptoms (≥1 symptom score ≥7);
  * Confirmed by clinicians.
Postoperative Rescue Treatment Medication Use | Within 6 months post-surgery.
  Record rescue treatment (oral methylprednisolone: days 1-5: 30 mg, days 6-10: 20 mg, days 11-15: 10 mg, days 16-20: 5 mg) initiation for symptom/polyp recurrence.
Postoperative Complications | Within 6 months after surgery.
  Record postoperative complications, including bleeding, infection, and altered Sense of Smell.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China